CLINICAL TRIAL: NCT06066164
Title: Cortical Excitability Among Substance Use Disorder Patients
Brief Title: Transcranial Magnetic Stimulation in Substance Use Disorder Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Goda, AbdGoda, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Tms in SUD patients
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator)
  Interventions: Device: Transcranial magnetic stimulation (TMS)
- Polysubstance use disorder patients (Active Comparator)
  Interventions: Device: Transcranial magnetic stimulation (TMS)
- Monosubstance use disorder patients (Active Comparator)
  Interventions: Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — Trans-cranial magnetic stimulation (TMS) is a safe and painless technique for evoking activity in neurons in the human brain through the intact scalp and skull To measure cortical excitability

SUMMARY:
To determine the effect of substance use disorder on cortical excitability using transcranial magnetic stimulation (TMS) , it's a scientific study

DETAILED DESCRIPTION:
The numbers for substance use disorders are large, and we need to pay attention to them. Data from the 2018 National Survey on Drug Use and Health suggest that, over the preceding year, 20.3 million people age 12 or older had substance use disorders, and 14.8 million of these cases were attributed to alcohol. When considering other substances, the report estimated that 4.4 million individuals had a marijuana use disorder and that 2 million people suffered from an opiate use disorder. It is well known that stress is associated with an increase in the use of alcohol and other substances, and this is particularly relevant today in relation to the chronic uncertainty and distress associated with the COVID-19 pandemic along with the traumatic effects of racism and social injustice,Trans-cranial magnetic stimulation (TMS) is a safe and painless technique for evoking activity in neurons in the human brain through the intact scalp and skull). Since its introduction in the mid-1980s is used to evaluate the cortico-spinal tract, cortical motor areas,, map motor and cognitive functions, study neural networks, and modulate brain function with a potential therapeutic aim, On one hand, the development of specific stimulation protocols, such as the cortical silent period (CSP) and paired-pulse paradigms, as well as the emerging concept that motor cortical output is affected by non-primary motor areas, including the ventral and dorsal premotor cortex, supplementary motor area, and cingulate cortex, has allowed the use of TMS to explore inhibitory and excitatory interactions within motor cortical regions in several neuropsychiatric disorders. Different TMS protocols can be used to study different components of cortical excitability and provide insight in to the regulation of different neurotransmitter systems.

ELIGIBILITY:
Inclusion Criteria:

1. Age:above18yearsold
2. males only
3. Patients fulfilling diagnostic criteria of substance use disorder according to DSM-5

Exclusion Criteria:

* 1. patients with other comorbid psychatric disorders. 2-patients with medical disease. 3.patients wirh epilepsy or family history of epilepsy. 4-cardiac pacemaker 5-metal implants in head as participant will be applied to magnetic field of the TMS 6-age yonnger than 18

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Measure cortical excitability in substance use disorder patients by TMS | Baseline
  Estimation of cortical excitability in substance use disorder patients and compare it in mono substance use disorder patients and poly substance use disorder patients

IPD SHARING:
Plan to Share IPD: Yes